CLINICAL TRIAL: NCT07291661
Title: The Role of Anorectal Manometry in Diagnosing and Guiding Management of Pediatric Chronic Refractory Constipation
Brief Title: The Role of Anorectal Manometry in Pediatric Chronic Refractory Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abd Elaal Ahmed, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Anorectal manometry
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Refractory Constipation; Fecal Incontinence in Children
Keywords: Anorectal manometry; Functional constipation; Pediatric chronic refractory constipation; Fecal incontinence; Biofeedback therapy; Botox injection
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: A descriptive cross-sectional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High resolution anorectal manometry using multiuse water perfused catheter (Other): Solar™ GI High Resolution Anorectal Manometry with multiuse water perfused catheter
  Interventions: Device: High resolution anorectal manometry using a multiuse water perfused catheter

INTERVENTIONS:
Device: High resolution anorectal manometry using a multiuse water perfused catheter — According to the international anorectal physiology working group recommendations(8):
  Stabilization: A 3-minute period after catheter insertion to allow anal tone to return to baseline.
  * Rest: Measures basal anal tone over 60 seconds.
  * Squeeze: Records anal pressure during voluntary contraction. Three 5-second squeezes are performed.
  * Long Squeeze: Evaluates anal pressure and fatigue during a single sustained 30-second contraction.
  * Cough: Assesses reflex anal pressure changes during two single coughs.
  * Push: Measures pressure changes during simulated defecation. Three 15-second pushes are performed.
  * RAIR (Rectoanal Inhibitory Reflex): Tests reflex anal relaxation after rapid rectal balloon distension, starting with at least 30 mL.
  Rectal Sensory Test: Measures rectal sensitivity by recording balloon volumes at three thresholds: first constant sensation, desire to defecate, and maximum tolerated volumes.
  · Balloon Expulsion: time required to expel the balloon.

SUMMARY:
This research protocol outlines a two-year descriptive cross-sectional study to investigate the role of high-resolution anorectal manometry (HRAM) in children aged 4-18 years with chronic refractory constipation.The study plans to enroll 54 patients at Ain Shams University Specialized Hospital . The study aims to identify different patterns of anorectal dysfunction (like dyssynergic defecation or rectal hyposensitivity) using standardized international protocols. A key goal is to determine if these manometry findings can directly guide specific management strategies, such as biofeedback therapy for dyssynergia or botulinum toxin injections for anal hypertension. improving outcomes for children who do not respond to standard constipation therapies.

DETAILED DESCRIPTION:
Structural and functional abnormalities of the anorectum or pelvic floor have been observed in constipated children with or without fecal incontinence. Childhood functional constipation accounts for about 95% of cases, while organic causes are less than 5%.

Organic causes include Hirschsprung disease, anorectal malformations, neuromuscular disorders and metabolic causes. Functional constipation can be caused by paradoxical contraction or insufficient relaxation of the pelvic floor muscles, and/or inadequate rectal propulsive forces during defecation. According to the Rome IV criteria, functional constipation is defined separately for infants and toddlers (<4 years) and for children (≥ 4 years).

Anorectal manometry (ARM) is an objective tool used to measure pressure and sensation in the anorectum at rest, during squeezing, and during simulated evacuation. three dimensional high resolution anorectal manometry (3D-HRAM) employs an array of 256 sensors, offering a more detailed assessment of anorectal anatomy and function.

Anorectal manometry is used for the evaluation of chronic constipation by checking rectoanal coordination and rectal sensitivity, and helps exclude structural disorders. It evaluates fecal incontinence by analyzing sphincter function and rectal sensation, identifies sphincter hypertension in functional anorectal pain, and provides preoperative baseline data before surgeries affecting continence or defecation.

Treatment of childhood constipation includes both nonpharmacological approaches (education, dietary modifications, behavioral strategies, biofeedback, and pelvic floor physiotherapy) and pharmacological options (osmotic and stimulant laxatives, probiotics as well as newer medications such as prucalopride and lubiprostone). For children with persistent constipation transanal irrigation, botulinum toxin injections, neuromodulation, and surgical procedures may be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged from 4 to 18 years.
2. Participants who have chronic refractory constipation either functional or organic with or without fecal incontinence.
3. Cooperative patients.

Exclusion Criteria:

1. Children aged less than 4 years old.
2. Uncooperative patients.
3. Children with anal fissures or any painful conditions that interfere with the procedure.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of anorectal manometry abnormalities in children with chronic refractory constipation, with or without fecal incontinence. | Baseline
  We will measure resting anal pressure, squeeze pressure, changes in rectoanal pressure during cough and during stimulated defecation, rectoanal inhibitory reflex (RAIR), and rectal sensation thresholds (first sensation, urge, maximum tolerable volume) using High resolusion anorectal manometry(HRAM) .
  Abnormalities will be categorized as:
  * Impaired or absent RAIR
  * Abnormal resting or squeeze sphincter pressure (outside age-adjusted norms)
  * Rectal sensory dysfunction (hyposensitivity or hypersensitivity)
  * Presence of dyssynergic defecation. And will be reported as counts and percentages.

SECONDARY OUTCOMES:
Guiding Management of Chronic Refractory Constipation in Children Using Anorectal Manometry Findings. | Baseline
  Classification of anorectal manometry patterns-including dyssynergic defecation, rectal hyposensitivity, and elevated resting anal sphincter pressure-and documentation of the number of participants assigned to different management strategies including (biofeedback therapy, botulinum toxin injection) according to these findings.
  Patients with manometry parameters showing dyssennergic defecation or rectal hyposensitivity will receive biofeedback sessions. While Participants with manometry parameters showing high anal canal resting pressure will have botulinium toxin injections.

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa H. Ibrahim, Professor, Study Director — Assiut University- Faculty of medicine; Naglaa S. Mohamed, A. professor, Study Chair — Assiut University- Faculty of medicine; Rehab I. Hassan, Lecturer, Study Chair — Assiut University- Faculty of medicine
Locations (1):
- Assiut University-faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poojari VS, Mirani S, Shetty NS, Shah I. Evaluation of constipation in children using high-resolution anorectal manometry. Trop Doct. 2021 Oct;51(4):527-531. doi: 10.1177/00494755211030362. Epub 2021 Jul 16. PMID 34270377
- [Background] Rao SSC, Tetangco EP. Anorectal Disorders: An Update. J Clin Gastroenterol. 2020 Aug;54(7):606-613. doi: 10.1097/MCG.0000000000001348. PMID 32692116
- [Background] Carrington EV, Scott SM, Bharucha A, Mion F, Remes-Troche JM, Malcolm A, Heinrich H, Fox M, Rao SS; International Anorectal Physiology Working Group and the International Working Group for Disorders of Gastrointestinal Motility and Function. Expert consensus document: Advances in the evaluation of anorectal function. Nat Rev Gastroenterol Hepatol. 2018 May;15(5):309-323. doi: 10.1038/nrgastro.2018.27. Epub 2018 Apr 11. PMID 29636555
- [Background] Koppen IJN, Vriesman MH, Saps M, Rajindrajith S, Shi X, van Etten-Jamaludin FS, Di Lorenzo C, Benninga MA, Tabbers MM. Prevalence of Functional Defecation Disorders in Children: A Systematic Review and Meta-Analysis. J Pediatr. 2018 Jul;198:121-130.e6. doi: 10.1016/j.jpeds.2018.02.029. Epub 2018 Apr 12. PMID 29656863